CLINICAL TRIAL: NCT00157937
Title: A Randomized, Open Label, Cross-Over Study Comparing Effectiveness for the Montelukast Sodium With Comparator in Mild to Moderate Persistent Asthmatics
Brief Title: A Study to Compare Effectiveness of Montelukast Sodium With Comparator in Mild to Moderate Persistent Asthmatics (0476-329)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0476-329; 2005_069
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-01

CONDITIONS: Asthma; Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic | interventions — montelukast; Duration of Therapy

INTERVENTIONS:
Drug: MK0476; montelukast sodium/Duration of Treatment: 16 weeks
Drug: Comparator: theophylline ER/Duration of Treatment: 16 weeks

SUMMARY:
Subjects have 8-week with montelukast sodium or comparator drug administration period, 2-week wash-out period and 8-week comparator drug or the drug administration period (with cross-over design) for assessment of the drug efficacy, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 60 with mild to moderate asthma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2003-02; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
FEV1

SECONDARY OUTCOMES:
AM-PEFR; daytime symptom score; treatment frequency of beta agonist; global assessment investigator's symptom assessment; Quality of Life Questionnaire for Adult Korean Asthmatics; QLQAKA

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC